CLINICAL TRIAL: NCT03939026
Title: A Single-Arm, Open-Label, Phase 1 Study Evaluating the Safety, Efficacy, and Cellular Kinetics/Pharmacodynamics of ALLO-501, an Anti-CD19 Allogeneic CAR T Cell Therapy, And ALLO-647, An Anti-CD52 Monoclonal Antibody, in Patients With Relapsed/Refractory Large B-Cell Lymphoma or Follicular Lymphoma
Brief Title: Safety and Efficacy of ALLO-501 Anti-CD19 Allogeneic CAR T Cells in Adults With Relapsed/Refractory Large B Cell or Follicular Lymphoma
Acronym: ALPHA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allogene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-501-201
Record Dates: First submitted 2019-04-04; First posted 2019-05-06 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory Large B Cell Lymphoma; Relapsed/Refractory Follicular Lymphoma
Keywords: CAR T; Cell Therapy; Allogeneic Cell Therapy; Cellular Immuno-therapy; AlloCAR T; ALLO-501; ALLO-647; LBCL; Lymphoma; Follicular Lymphoma; Large B-Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Follicular; Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALLO-647, ALLO-501 (Experimental)
  Interventions: Genetic: ALLO-501; Biological: ALLO-647; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: ALLO-501 — ALLO-501 is an allogeneic CAR T cell therapy targeting CD19
Biological: ALLO-647 — ALLO-647 is a monoclonal antibody that recognizes a CD52 antigen
Drug: Fludarabine — Chemotherapy for lymphodepletion
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion

SUMMARY:
The purpose of the ALPHA study is to assess the safety, efficacy, cell kinetics and immunogenicity of ALLO-501 in adults with relapsed or refractory large B-cell lymphoma or follicular lymphoma after a lymphodepletion regimen comprising fludarabine, cyclophosphamide, and ALLO-647.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of Large B-cell Lymphoma (LBCL) or Follicular Lymphoma.
* Relapse or refractory disease after at least 2 lines of chemotherapy
* At least 1 measurable lesion at time of screening.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Adequate hematological, renal, liver, pulmonary, and cardiac functions.

Exclusion Criteria:

* Current or history of central nervous system (CNS) lymphoma.
* Clinically significant CNS dysfunction.
* ASCT within last 6 weeks or allogeneic HSCT within last 3 months prior to ALLO-647.
* Prior treatment with anti-CD19 therapy, any gene therapy, any genetically modified cell therapy or adoptive T cell therapy
* Systemic anticancer therapy within 2 weeks prior to study entry.
* On-going treatment with immunosuppressive agents.
* Active acute or chronic graft versus host disease (GvHD), or GvHD requiring immunosuppressive treatment within 4 weeks of enrollment.
* Any form of primary or acquired immunodeficiency (e.g., severe combined immunodeficiency disease).
* Current thyroid disorder (including hyperthyroidism), except for subjects with hypothyroidism controlled on a stable dose of hormone replacement therapy.
* Patients unwilling to participate in an extended safety monitoring period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects experiencing Dose Limiting Toxicities at increasing doses of ALLO-501 | 28 days
  Dose limiting toxicity is defined as protocol-defined ALLO-501-related adverse events with onset within 28 days following infusion
Proportion of patients experiencing Dose Limiting Toxicity with ALLO-647 in combination with fludarabine/cyclophosphamide administered prior to ALLO-501 | 33 days
  Dose-limiting toxicity is defined as protocol-defined ALLO-647-related adverse events with onset within 33 days following 1st infusion

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Stanford University, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - St. Davids South Austin Medical Center, Austin, Texas
  - MD Anderson, Houston, Texas

REFERENCES:
- [Derived] Locke FL, Munoz JL, Tees MT, Lekakis LJ, de Vos S, Nath R, Stevens DA, Malik SA, Shouse GP, Hamadani M, Oluwole OO, Perales MA, Miklos DB, Fisher PW, Feng A, Navale L, Le Gall JB, Neelapu SS. Allogeneic Chimeric Antigen Receptor T-Cell Products Cemacabtagene Ansegedleucel/ALLO-501 in Relapsed/Refractory Large B-Cell Lymphoma: Phase I Experience From the ALPHA2/ALPHA Clinical Studies. J Clin Oncol. 2025 May 10;43(14):1695-1705. doi: 10.1200/JCO-24-01933. Epub 2025 Feb 13. PMID 39946666